CLINICAL TRIAL: NCT06749821
Title: The Acute Effect of Kinesio Tape on Pain, Joint Range of Motion and Dynamic Balance in Patients With Low Back Pain: Randomized Placebo-Controlled Trial
Brief Title: The Acute Effect of Kinesio Tape on Pain, Joint Range of Motion and Dynamic Balance in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Ilayda Dilan Isik, MsC Physiotherapist, Baskent University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: BaskentUni
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Low Back Pain
Keywords: Kinesio Tape; Low Back Pain; Balance; Joint Range of Motion
MeSH Terms: conditions — Low Back Pain | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio Tape Group (Active Comparator): Kinesio tape was applied to this group.
  Interventions: Other: Kinesio Tape
- Placebo Tape Group (Placebo Comparator): Placebo tape was applied to this group.
  Interventions: Other: Placebo Tape (Arm 1)
- Control Group (Other): No application was made to this group. Just rest
  Interventions: Other: Control (no last irrigation)

INTERVENTIONS:
Other: Kinesio Tape — Kinesio tape (KT) is an elastic therapeutic tape used to treat sports injuries and various other disorders. It was first used by Dr. Kenzo Kase in 1979 to relieve pain and promote healing in soft tissues and is a method that is constantly being updated. The KT method is a therapeutic taping technique that relieves pain and facilitates lymphatic drainage by microscopically lifting the skin.
  Arms: Kinesio Tape Group
Other: Placebo Tape (Arm 1) — In this application, taping was applied in the same way but with a plaster tape.
  Arms: Placebo Tape Group
Other: Control (no last irrigation) — No application was made.
  Arms: Control Group

SUMMARY:
The aim of this study is to evaluate the acute effect of kinesio taping on pain, range of motion and dynamic balance in patients with chronic nonspecific low back pain. 48 patients were included in the study and were randomly divided into three groups by ordinal number randomization. All patients were evaluated of pain, joint range of motion and dynamic balance before and 45 minutes after the application. Kinesio taping with elastic therapeutic tape was applied to the core muscles of the study group, and the same muscles of the placebo group were taped with plaster tape in the same way, and no application was made to the control group.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the acute effect of kinesio taping on pain, range of motion and dynamic balance in patients with chronic nonspecific low back pain. 48 patients were included in the study and were randomly divided into three groups by ordinal number randomization. All patients were evaluated by the same physiotherapist in terms of pain (Visual Analog Scale), joint range of motion (Gonyometric measurement) and dynamic balance (Timed Up and Go Test) before and 45 minutes after the application. Kinesio taping with elastic therapeutic tape was applied to the transversus abdominis, rectus abdominis and iliocostal muscles of the study group, and the same muscles of the placebo group were taped with plaster tape in the same way, and no application was made to the control group.

ELIGIBILITY:
Inclusion criteria for the study:

* Having low back pain of at least 3 out of 10 points on the Visual Analog Scale,
* Being between the ages of 30-55,
* Having low back pain for at least 3 months,
* Having been tested with a test piece beforehand and not having an allergy to kinesio taping.

Exclusion criteria for the study:

* Having had surgery for low back pain,
* Not complying with treatment,
* Having a neurological deficit,
* Being pregnant,
* Having received any treatment for low back pain in the last month.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 45 minute
  It will evaluate pain. People marked the severity of their pain on a 10 cm line. (0: no pain, 10: maximum pain) Pain was evaluated separately as activity, rest and night.
Goniometer | 45 minute
  Joint range of motion was measured with a goniometer. Spinal flexion, extension and lateral flexion were evaluated.
Timed up and go test | 45 minute
  Dynamic balance was assessed with timed get up and go. The person stood up from a fixed chair, walked 3 meters and sat back down, and the time spent during this time was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Animarapha Manual Therapy and Reflexology Center, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Shareef AT, Omar MTA, Ibrahim AHM. Effect of Kinesio Taping on Pain and Functional Disability in Chronic Nonspecific Low Back Pain: A Randomized Clinical Trial. Spine (Phila Pa 1976). 2016 Jul 15;41(14):E821-E828. doi: 10.1097/BRS.0000000000001447. PMID 27392262